CLINICAL TRIAL: NCT02459275
Title: PEP uP Protocol (Enhanced Protein-Energy Provision Via the Enteral roUte Feeding Protocol) in Surgical Patients
Brief Title: PEP uP Protocol in Surgical Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding discontinued
Sponsor: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Collaborators: Nestle Health Science (Industry)
Responsible Party: Principal Investigator, Daniel D Yeh, MD, Daniel Dante Yeh, MD, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PEP uP Surgical RCT
Record Dates: First submitted 2015-05-27; First posted 2015-06-02 (Estimated); Results first posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Critically Ill
Keywords: feeding protocol; enteral nutrition protocol; critically ill; surgical ICU; enteral nutrition; nutrition therapy
MeSH Terms: conditions — Critical Illness | interventions — Metoclopramide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEP uP Protocol (Experimental): Participants will receive the PEP uP protocol with the pro motility agent. The intervention will be provided until the tube feeds are stopped or patient is fed meals orally and will be tracked until hospital discharge or 60 days which ever occur first.
  Interventions: Other: PEP uP Protocol; Drug: Metoclopramide
- Standard of Care (No Intervention): Standard formula polymeric tube feeds started at a rate of 20 ml/hour. Gastric residual volume (GRV) will be checked every 4 hours. GRV is reinfused to the patient each time it is checked. GRV threshold is 200-500 ml. If the patient is tolerating tube feeds as determined by measuring the GRV, the rate is advanced by 20 ml/hour every 4 hours up to the goal rate. Participants will be followed until the tube feeds are stopped or patient is fed meals orally and will be tracked until hospital discharge or 60 days which ever occur first.

INTERVENTIONS:
Other: PEP uP Protocol — Semi-elemental tube feeds are started at the hourly goal rate as determined by the 24 hour volume goal. Protein supplements will be started at the initiation of tube feeds to target a daily delivery of 2 g/kg/day.
  Arms: PEP uP Protocol
Drug: Metoclopramide — Metoclopramide 10mg Intravenous (IV) every 6 hours (q6h) or 5mg IV q6h for renal failure will be started empirically concomitant with EN initiation. Gastric Residual Volume (GRV) will be checked every 4 hours and will be reinfused to the patient each time it is checked.
  Other Names: Reglan
  Arms: PEP uP Protocol

SUMMARY:
The main objective of this project is to asses for safety, feasibility and effectiveness of an aggressive feeding protocol, PEP uP (Enhanced Protein-Energy Provision via the Enteral Route Feeding Protocol) in increasing protein and energy delivery to critically ill surgical patients. Our hypothesis is that an aggressive feeding protocol, PEP uP will be safe, acceptable, and effectively increase protein and energy delivery to critically ill surgical patients.

DETAILED DESCRIPTION:
Gross underfeeding or iatrogenic malnutrition is prevalent in intensive care units throughout the world. Critically ill patients only receive, on average, 40-50% of their prescribed nutritional requirements. Inadequate provision of nutrition to these patients is associated with increased complications, prolonged length of stay in the ICU and hospital, and increased mortality. There are good data from large scale observational studies and randomized trials that suggest better fed patients have better clinical and economic outcomes and there are ICUs that consistently reach an average of 80-90% nutritional adequacy (amount of nutrition received over amount prescribed) thus it appears to be a feasible goal.

The PEP uP protocol (Enhanced Protein-Energy Provision via the Enteral Route Feeding Protocol) includes a new, innovative approach that protocolizes an aggressive set of strategies to providing enteral nutrition (EN) and shifts the paradigm from reactionary to proactive followed by de-escalation if nutrition therapy is not needed. The key components of this new PEP uP protocol are the following:

1. Starting feeds at the target rate based on increasing evidence that some patients tolerate starting nutrition at a higher rate of delivery and that slow start ups are not necessary.
2. Allowing "trophic feeds" a low volume of a concentrated feeding solution for 24 hours or longer, designed to maintain gastrointestinal structure and function for those patients who are deemed unsuitable for high volume intragastric feeds.
3. Prescribing semi-elemental feeding solution instead of a standard polymeric solution.

   These can then be changed to more traditional polymeric solution once the patient is tolerating adequate amounts of nutrition.
4. Prescribing protein supplements at initiation of EN and then discontinue if EN is well tolerated and protein requirement are met through their standard EN.
5. Starting motility agents at the same time EN is started with a re-evaluation in the days following to see if it is necessary.

This PEP uP protocol has been previously studied in two published studies enrolling primarily medical patients. In the first study, a pilot before and after trial, the protocol seemed to be feasible, safe, and acceptable to critical care nurses. No incidents compromising patient safety were observed. (Heyland 2010) Rates of vomiting, regurgitation, aspiration, and pneumonia were similar and the PEP uP group received significantly more energy and protein (when they were prescribed to receive full volume as opposed to "trophic"). A subsequent multi-center cluster randomized trial involving low-performing ICUs likewise demonstrated that intervention sites had improvements in energy and protein delivery as well as a decrease in average time from ICU admission to start of enteral nutrition compared to the control group. (Heyland 2013).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ICU admission within past 48 hours
* Initiation of tube feeds currently planned by the surgical ICU (SICU) team and primary surgical team
* Admitted by a surgical service to the SICU (not a medical ICU or neurology patient)
* Expected to remain mechanically ventilated for > 24 h and expected to require ICU care for > 72 h after screening

Exclusion Criteria:

* Pregnancy
* Attending surgeon preference (they must agree to feeding their patient according to the protocol in either arm using the goal rate determined by the SICU team and the nutritionist)
* Contraindication to enteral nutrition (bowel obstruction, bowel discontinuity, proximal enterocutaneous fistula, and short gut syndrome)
* Do not resuscitate (DNR) status or goals of care that specify limitations in medical therapies
* Death expected within 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-07; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daren K Heyland, MD, Study Director — Clinical Evaluation Research Unit
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Jamaica Hospital Medical Center, Jamaica, New York
  - Virginia Tech Carilion School of Medicine, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heyland DK, Cahill NE, Dhaliwal R, Wang M, Day AG, Alenzi A, Aris F, Muscedere J, Drover JW, McClave SA. Enhanced protein-energy provision via the enteral route in critically ill patients: a single center feasibility trial of the PEP uP protocol. Crit Care. 2010;14(2):R78. doi: 10.1186/cc8991. Epub 2010 Apr 29. PMID 20429886
- [Background] Heyland DK, Murch L, Cahill N, McCall M, Muscedere J, Stelfox HT, Bray T, Tanguay T, Jiang X, Day AG. Enhanced protein-energy provision via the enteral route feeding protocol in critically ill patients: results of a cluster randomized trial. Crit Care Med. 2013 Dec;41(12):2743-53. doi: 10.1097/CCM.0b013e31829efef5. PMID 23982032
- [Background] Heyland DK, Dhaliwal R, Lemieux M, Wang M, Day AG. Implementing the PEP uP Protocol in Critical Care Units in Canada: Results of a Multicenter, Quality Improvement Study. JPEN J Parenter Enteral Nutr. 2015 Aug;39(6):698-706. doi: 10.1177/0148607114531787. Epub 2014 Apr 18. PMID 24748597
- [Background] McCall M, Cahill N, Murch L, Sinuff T, Bray T, Tanguay T, Heyland DK. Lessons Learned From Implementing a Novel Feeding Protocol: Results of a Multicenter Evaluation of Educational Strategies. Nutr Clin Pract. 2014 Aug;29(4):510-517. doi: 10.1177/0884533614531047. Epub 2014 Apr 22. PMID 24757062
- See also: Critical Care Nutrition website including information on the PEP uP Protocol — http://www.criticalcarenutrition.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PEP uP Protocol | Standard of Care
Started | 19 | 17
Completed | 19 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEP uP Protocol | Standard of Care | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.1 (24.7) | 50.6 (15.6) | 49.8 (0.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 18 | 12 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Total Amount of Protein Received
Description: The total amount of protein received from either EN or parenteral nutrition (PN), inclusive of propofol, divided by the amount prescribed as per the baseline assessment and expressed as a percentage.
Time Frame: 12 days
Measure: Mean (Standard Deviation); unit: percentage of protein
Arm/Group | PEP uP Protocol | Standard of Care
Number analyzed (Participants) | 19 | 17
percentage of protein | 55.1 (24.4) | 52.9 (23.2)

2. Primary Outcome: Total Amount of Energy
Description: The total amount of energy received from either EN or parenteral nutrition (PN), inclusive of propofol, divided by the amount prescribed as per the baseline assessment and expressed as a percentage.
Time Frame: 12 days
Measure: Mean (Standard Deviation); unit: percentage of energy
Arm/Group | PEP uP Protocol | Standard of Care
Number analyzed (Participants) | 19 | 17
percentage of energy | 49.4 (23.7) | 60.3 (22.8)

3. Secondary Outcome: Time to Initiation of Enteral Nutrition
Description: Hours from intensive care unit (ICU) admission
Time Frame: 12 days
Measure: Mean (Inter-Quartile Range); unit: hours
Arm/Group | PEP uP Protocol | Standard of Care
Number analyzed (Participants) | 19 | 17
hours | 26.7 [20 to 37.5] | 28.2 [22.3 to 33.5]

4. Secondary Outcome: ICU Length of Stay
Description: Days in the intensive care unit
Time Frame: up to 60 days
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | PEP uP Protocol | Standard of Care
Number analyzed (Participants) | 19 | 17
days | 12 [6 to 41.7] | 12.5 [10.6 to 15.9]

5. Secondary Outcome: Mortality
Description: Number of participants that died
Time Frame: up to 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | PEP uP Protocol | Standard of Care
Number analyzed (Participants) | 19 | 17
Participants | 1 | 2

6. Secondary Outcome: Hospital Length of Stay
Description: Days the participants were in the admitted in the hospital
Time Frame: up to 60 days
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | PEP uP Protocol | Standard of Care
Number analyzed (Participants) | 19 | 17
days | 21.4 [14.9 to 60] | 16.6 [13.9 to 21.1]

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | PEP uP Protocol | Standard of Care
All-Cause Mortality (participants affected / at risk) | 1/19 | 2/17
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/17
Other Adverse Events (participants affected / at risk) | 0/19 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEP uP Protocol (N=19) | Standard of Care (N=17)
temporary QTC prolongation (Cardiac disorders) | 1 (1) | 0 (0) — temporary QTC prolongation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT02459275/Prot_SAP_000.pdf